CLINICAL TRIAL: NCT02069041
Title: Phase 1b Study of 5-FU/FA and Oxaliplatin (FOLFOX4) Plus Ramucirumab (LY3009806) in Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Study of Ramucirumab (LY3009806) in Participants With Advanced Liver Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15233; I4T-CR-JVCQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-02-20; First posted 2014-02-21 (Estimated); Results first posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2017-09

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Ramucirumab; Folfox protocol; Leucovorin; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ramucirumab + FOLFOX4 (Experimental): 8 milligram/kilogram (mg/kg) ramucirumab given intravenously (IV) on Day 1 followed by FOLFOX4 (folinic acid + fluorouracil + oxaliplatin chemotherapy regimen) given IV on Day 1 of 2 week cycles:
  FOLFOX4 every 2 weeks:
  85 milligram per square meter (mg/m²) oxaliplatin IV on Day 1 200 mg/m² folinic acid(FA) IV on days 1 and 2 400 mg/m² 5-FU bolus on days 1 and 2 600 mg/m2 5-FU 22-h continuous infusion on Days 1 and 2
  Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Biological: Ramucirumab; Drug: FOLFOX4

INTERVENTIONS:
Biological: Ramucirumab — Administered IV.
  Other Names: IMC-1121B; LY3009806
Drug: FOLFOX4 — Administered IV.
  Other Names: FOLFOX4 (leucovorin + fluorouracil + oxaliplatin)

SUMMARY:
The main purpose of this study is to determine if the advised dose of ramucirumab is safe to be taken with chemotherapy treatment in participants with advanced liver tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of hepatocellular carcinoma (HCC) or imaging findings consistent with HCC in a participant with liver cirrhosis and alpha-fetoprotein > 200 nanogram per milliliter
* At least 1 measurable or non-measurable lesion
* Child-Pugh A
* Barcelona Clinic Liver Cancer (BCLC) stage C or BCLC stage B not amenable to locoregional therapy or refractory to locoregional therapy
* Eastern Cooperative Oncology Group Performance Status of 0 or 1
* Have not received previous systemic therapy for advanced HCC
* Have resolution to Grade ≤1 of all clinically significant toxic effects of prior locoregional therapy
* Adequate organ function including: Absolute neutrophil coun t≥1.5×109/liter (L), hemoglobin ≥9 gram/deciliter, and platelets ≥90×109/L; Total bilirubin level ≤1.5 the upper limit of the normal range (ULN), aspartate transaminase and alanine transaminase ≤5 ULN, albumin >28 gram/L; Serum creatinine level ≤1.5 ULN; or calculated serum creatinine clearance ≥50 milliliter/minute; International Normalized Ratio≤1.5 and partial thromboplastin time ≤5 seconds above ULN
* The urinary protein is ≤ 1+. If ≥ 2+ proteinuria, the 24-hour urine protein is <1000 milligram
* An estimated life expectancy of at least 12 weeks

Exclusion Criteria:

* Received any investigational therapy or non-approved drug within 28 days prior to enrollment
* Undergone major surgery within 28 days prior to enrollment, or undergone central venous access device placement within 7 days prior to enrollment
* Undergone hepatic locoregional therapy within 28 days prior to enrollment
* Undergone radiation to any nonhepatic site within 14 days prior to enrollment
* Prior liver transplant
* Fibrolamellar carcinoma or cholangiocellular carcinoma
* Received any transfusion, blood component preparation, erythropoietin, albumin preparation, or granulocyte-colony stimulating factors within 14 days prior to enrollment
* Receiving therapeutic anticoagulation with warfarin, low-molecular weight heparin, or similar agents
* Receiving ongoing therapy with nonsteroidal anti-inflammatory agents or other antiplatelet agents.
* Known human immunodeficiency virus infection or acquired immunodeficiency syndrome-related illness
* Active or uncontrolled clinically serious infection
* Uncontrolled thrombotic or hemorrhagic disorder
* Serious or nonhealing wound, ulcer, or bone fracture within 28 days prior to enrollment
* History of gastrointestinal perforation or obstruction
* History of or current hepatic encephalopathy or current clinically meaningful ascites
* Known allergy to monoclonal antibody, fluorouracil, oxaliplatin or their excipients
* Interstitial pneumonia or interstitial fibrosis of the lung
* Central nervous system metastases or carcinomatous meningitis
* Known history of dihydropyrimidine dehydrogenase deficiency
* Symptomatic congestive heart failure, unstable angina pectoris, or symptomatic or poorly controlled cardiac arrhythmia
* Experienced any arterial thromboembolic event
* Uncontrolled arterial hypertension
* Grade 3-4 venous thromboembolic events occurring within 3 months prior to enrollment
* Experienced any grade 3-4 gastrointestinal bleeding or any variceal bleeding episode in the 3 months prior to enrollment requiring transfusion, endoscopic or operative intervention
* Esophageal or gastric varices that require immediate intervention or represent a high bleeding risk
* Pre-existing grade ≥ 2 motor or sensory neuropathy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taoyuan

REFERENCES:
- [Derived] Lin CC, Yang TS, Yen CJ, Cheng R, Liu J, Hsu C. Safety and Preliminary Efficacy of Ramucirumab in Combination with FOLFOX4 in Patients with Advanced Hepatocellular Carcinoma: A Nonrandomized, Open-Label, Phase Ib Study. Oncologist. 2020 Dec;25(12):e1921-e1929. doi: 10.1002/onco.13550. Epub 2020 Oct 31. PMID 33017497

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants completed the study if they completed 3 cycles or discontinued due to a DLT during the DLT assessment period.
Period: Overall Study
Arm/Group | Ramucirumab + FOLFOX4
Started | 8
Received at Least One Dose of Study Drug | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Arm/Group | Ramucirumab + FOLFOX4
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.56 (11.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 8
Basis of Initial Pathological Diagnosis [Count of Participants; unit: Participants] — Population: All participants who received at least one dose of study drug and had baseline initial pathological diagnosis data.
  Participants
    Histopathological: number analyzed (Participants) | 6
    Histopathological | 3
    Cytological: number analyzed (Participants) | 6
    Cytological | 1
    Biochemical Assay and Imaging: number analyzed (Participants) | 6
    Biochemical Assay and Imaging | 2
Disease Stage [Count of Participants; unit: Participants] — Stage means how big the tumor is and how far it has spread. Stages range from I (spread to nearby tissue) to IV (spread throughout the body). Population: All participants who received at least one dose of study drug and had baseline disease stage data.
  Participants
    Stage I: number analyzed (Participants) | 6
    Stage I | 0
    Stage II: number analyzed (Participants) | 6
    Stage II | 1
    Stage III: number analyzed (Participants) | 6
    Stage III | 4
    Stage IV: number analyzed (Participants) | 6
    Stage IV | 1
    Unknown: number analyzed (Participants) | 6
    Unknown | 0
Duration of Disease (months) [Median (Full Range); unit: months] — Duration of disease is time from date of histology/cytologic confirmation of advanced solid tumor to date of first dose. Population: All participants who received at least one dose of study drug and had baseline duration of disease data.
  months
    number analyzed (Participants) | 6
    (all) | 0.345 [0.23 to 0.66]
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Following are ECOG grades. 0: Fully active, perform all pre-disease activities without restriction. 1: Restricted in physically strenuous activity but ambulatory, carry out work of a light or sedentary nature. 2: Ambulatory, capable of selfcare, unable to carry out any work activities, up and about more than (>) 50% of waking hours. 3: Capable of limited selfcare, confined to bed or chair >50% of waking hours. 4: Completely disabled, not capable of any selfcare, totally confined to bed or chair. 5: Dead. Participants in "Not reported" category were on study, had no data for this time point.
  Participants
    0 | 4
    1 | 4
    2 | 0
    >2 | 0
    Missing | 0
Barcelona Clinic Liver Cancer (BCLC) Classification [Count of Participants; unit: Participants] — The following is BCLC classification:
  Stage A: Early hepatocellular carcinoma. Stage B: Intermediate hepatocellular carcinoma. Stage C: Advanced hepatocellular carcinoma. Stage D: End stage hepatocellular carcinoma.
  Participants
    Stage A | 0
    Stage B | 1
    Stage C | 7
    Stage D | 0
    Missing | 0
Viral hepatitis B [Count of Participants; unit: Participants]
  Test Positive | 8
  Test Negative | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of other non-serious Adverse Events (AEs), and all Serious Adverse Events (SAE's), regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline through study completion (Up To 8 Months)
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ramucirumab + FOLFOX4
Number analyzed (Participants) | 8
Participants | 4

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Ramucirumab
Description: Maximum Concentration (Cmax)
Time Frame: Cycle 1 and Cycle 3: 0,1.0,1.5,2.0,3.0,5.0,24.0,48.0,168.0,336.0 hours
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL(microgram / milliliter)
Arm/Group | Ramucirumab + FOLFOX4
Number analyzed (Participants) | 8
ug/mL(microgram / milliliter)
  Cycle 1 | 155 (25)
  Cycle 3: number analyzed (Participants) | 3
  Cycle 3 | 190 (29)

3. Secondary Outcome: PK:Area Under the Concentration-Time Curve (AUC[0-∞]) of Ramucirumab
Description: Area under the concentration-time curve.
Time Frame: Cycle 1 and Cycle 3: 0,1.0,1.5,2.0,3.0,5.0,24.0,48.0,168.0,336.0 hours
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day / milliliter)(ug*day/mL)
Arm/Group | Ramucirumab + FOLFOX4
Number analyzed (Participants) | 8
microgram*day / milliliter)(ug*day/mL)
  Cycle 1: number analyzed (Participants) | 6
  Cycle 1 | 940 (24)
  Cycle 3: number analyzed (Participants) | 3
  Cycle 3 | 1190 (25)

4. Secondary Outcome: Number of Participants With Anti-Ramucirumab Antibodies
Time Frame: Baseline through 6.1 Months
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ramucirumab + FOLFOX4
Number analyzed (Participants) | 8
Participants | 0

5. Secondary Outcome: Percentage of Participants With Best Response of Complete Response (CR) or Partial Response (PR) (Overall Response Rate [ORR])
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST, version[v] 1.1) criteria.CR was defined as the disappearance of all target and non-target lesions and all target and non-target lymph nodes were non-pathological or normal in size [<10 millimeter (mm) short axis]. PR is at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters. Progressive Disease(PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (including the baseline sum if that is the smallest).In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
  Percentage of participants with CR or PR= (number of participants whose best overall response was CR or PR)/(number of participants treated)*100.
Time Frame: Response to Disease Progression or Death (Up To 7 Months)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of Participants
Arm/Group | Ramucirumab + FOLFOX4
Number analyzed (Participants) | 8
percentage of Participants | 25

ADVERSE EVENTS:
Description: All participants who received at least one dose of study drug.
Arm/Group | Ramucirumab + FOLFOX4
Serious Adverse Events (participants affected / at risk) | 5/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab + FOLFOX4 (N=8)
Ascites (Gastrointestinal disorders) | 2 (2)
Pyrexia (General disorders) | 3 (5)
Hepatic haemorrhage (Hepatobiliary disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2)
Neutrophil count decreased (Investigations) | 2 (2)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab + FOLFOX4 (N=8)
Anaemia (Blood and lymphatic system disorders) | 3 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 6 (10)
Abdominal pain upper (Gastrointestinal disorders) | 3 (6)
Ascites (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 5 (9)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (2)
Mouth ulceration (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 4 (7)
Stomatitis (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 2 (5)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (7)
Malaise (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 3 (4)
Pyrexia (General disorders) | 2 (8)
Influenza (Infections and infestations) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (2)
Alanine aminotransferase increased (Investigations) | 2 (5)
Aspartate aminotransferase increased (Investigations) | 2 (6)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (3)
Blood creatinine increased (Investigations) | 2 (4)
Gamma-glutamyltransferase increased (Investigations) | 1 (2)
Neutrophil count decreased (Investigations) | 5 (7)
Platelet count decreased (Investigations) | 4 (12)
Weight decreased (Investigations) | 2 (2)
Weight increased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 3 (9)
Decreased appetite (Metabolism and nutrition disorders) | 5 (9)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (10)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (3)
Dizziness (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (3)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (3)
Proteinuria (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (3)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days